CLINICAL TRIAL: NCT03177720
Title: Determination of Single-dose Intrapulmonary Pharmacokinetics of Ciprofloxacin and Imipenem in Healthy Subjects and Intubated Patients Suffering From Pneumonia Using Bronchoalveolar Lavage
Brief Title: Evaluation of Innovative Tools in Development of Antibiotics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Markus Zeitlinger, Professor Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ELF Cipro
Record Dates: First submitted 2017-05-30; First posted 2017-06-06 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Ciprofloxacin; Imipenem

STUDY DESIGN:
Intervention Model Description: 24 patients and 18 healthy volunteers are included. 12 patients and 9 volunteers are receiving imipenem as study drug, the other 12 patients and 9 volunteers receive ciprofloxacin.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofloxacin (Active Comparator): Half of patients and healthy volunteers are receiving ciprofloxacin, the other half imipenem.
  Interventions: Drug: Ciprofloxacin
- Imipenem (Active Comparator): Half of patients and healthy volunteers are receiving ciprofloxacin, the other half imipenem.
  Interventions: Drug: Imipenem

INTERVENTIONS:
Drug: Ciprofloxacin — Ciprofloxacin 400mg will be administered as single dose infusion over 60 minutes, imipenem/cilastatin 1000mg as single intravenous dose applicated over 60 minutes.
  Arms: Ciprofloxacin
Drug: Imipenem — Ciprofloxacin 400mg will be administered as single dose infusion over 60 minutes, imipenem/cilastatin 1000mg as single intravenous dose applicated over 60 minutes.
  Arms: Imipenem

SUMMARY:
The investigators will determine the difference of pharmacokinetics of ciprofloxacin and imipenem between healthy volunteers and intensive care patients suffering from pneumonia in plasma and at the target site - lung - using bronchoalveolar lavage. As additional aspect the feasibility of combining microdosing of C14 ciprofloxacin with microdialysis, saliva sampling and bronchoalveolar lavage is studied by comparing pharmacokinetics of microdose and macrodose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 55 years
* Good state of health (mentally and physically)
* Body mass index within a range of 18 to 28kg/m2 inclusive.
* Non-Smoker
* A signed and dated written informed consent form.
* The subject is able to understand and willing to comply with protocol requirements and timetables, instructions and protocol-stated restrictions.
* Negative serology (human immunodeficiency virus, hepatitis B-AG and C-AB) at screening.
* Vital signs should be within the following ranges:
* Oral or tympanic temperature between 35 and 37.5°C.
* Systolic blood pressure, 90-140 mmHg.
* Diastolic blood pressure, 50-90 mmHg.
* Pulse rate, 50-90 bpm.

Exclusion Criteria:

* Any acute or chronic illness or clinically relevant (Investigator's judgement) abnormality identified on the screening medical assessment, laboratory tests or ECG, unless in the opinion of the Investigator it will not interfere with the study procedures, affect the outcome of the study or compromise the safety of the subject.
* All subjects with known seizure disorder, with the exception of a febrile seizure in childhood
* Use of prescription or non-prescription drugs within 7 days or 10 times the elimination half-life (whichever is longer) prior to the first dose of study medication.
* Any intake of grapefruit juice within 1 week prior to the first dose.
* Allergies (except for mild forms of hay fever), a history of hypersensitivity reactions including psychological or neurological symptoms or signs, or anaphylactic shock following administration of any medicine.
* Allergy to or any contraindication against the active or inactive ingredients in the study medication (ciprofloxacin, imipenem, cilastatin, propofol, midazolam, remifentanil, xylocain, and sevoflurane) and radioactive labelling with 14C.
* Smoker
* Alcohol or drug abuse
* Participation in a trial with any drug within 30 days or five half-lives (whichever is longer) before the start of the study.
* Donation of blood within a period of 4 weeks prior to dosing.
* Creatinine clearance ≤70mL/min/1.73m3
* Any other reason that the Investigator considers to make the subject unsuitable to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05-29 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Cmax (peak concentration in plasma and epithelial lining fluid) of imipenem and ciprofloxacin | Plasma over 10 hours and BAL (bronchoalveolar lavage) Sampling at different time points in these 10 hours.
  Comparison of Cmax of ciprofloxacin and imipenem in plasma and epithelial lining fluid, alveolar macrophages and saliva (only healthy subjects) in healthy subjects and patients with bacterial pneumonia.
AUC (area under the concentration curve in plasma and epithelial lining fluid) of imipenem and ciprofloxacin. | Plasma over 10 hours and BAL Sampling at different time points in these 10 hours.
  Comparison of AUC of ciprofloxacin and imipenem in plasma and epithelial lining fluid, alveolar macrophages and saliva (only healthy subjects) in healthy subjects and patients with bacterial pneumonia.
Tmax (time of peak concentration in plasma and epithelial lining fluid) of imipenem and ciprofloxacin. | Plasma over 10 hours and BAL Sampling at different time points in these 10 hours.
  Comparison of AUC of ciprofloxacin and imipenem in plasma and epithelial lining fluid, alveolar macrophages and saliva (only healthy subjects) in healthy subjects and patients with bacterial pneumonia.
Cmax (peak concentration in plasma, epithelial lining fluid and microdialysate) of C14 ciprofloxacin (microdose) | Plasma sampling over 10 hours and microdialysate sampling.
  Comparison of pharmacokinetics of microdoses and macrodoses in lung, subcutaneous tissue (microdialysis) and plasma in healthy volunteers.
AUC (area under the curve in plasma, epithelial lining fluid and microdialysate) of C14 ciprofloxacin (carbon-14 radiolabelled compound, microdose) | Plasma sampling over 10 hours and microdialysate sampling.
  Comparison of pharmacokinetics of microdoses and macrodoses in lung, subcutaneous tissue (microdialysis) and plasma in healthy volunteers.
Tmax (time of peak concentration in plasma, epithelial lining fluid and microdialysate) of C14 ciprofloxacin (microdose) | Plasma sampling over 10 hours and microdialysate sampling.
  Comparison of pharmacokinetics of microdoses and macrodoses in lung, subcutaneous tissue (microdialysis) and plasma in healthy volunteers.
Cmax (peak concentration in microdialysate) of ciprofloxacin (macrodose) | Microdialysate sampling (Baseline sampling before study drug administration - sampling over 3 hours - retrodialysis)
  In healthy volunteers only for comparison of Cmax of C14 ciprofloxacin and Cmax of ciprofloxacin as macrodose.
AUC (area under the concentration curve in microdialysate) of ciprofloxacin (macrodose) | Microdialysate sampling (Baseline sampling before study drug administration - sampling over 3 hours - retrodialysis)
  In healthy volunteers only for comparison of Cmax of C14 ciprofloxacin and Cmax of ciprofloxacin as macrodose.
Tmax (time of peak concentration in microdialysate) of ciprofloxacin (macrodose) | Microdialysate sampling (Baseline sampling before study drug administration - sampling over 3 hours - retrodialysis)
  In healthy volunteers only for comparison of Cmax of C14 ciprofloxacin and Cmax of ciprofloxacin as macrodose.

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | Screening visit and final examination are performed up to 7 days before/after the actual study day and safety and tolerability assessed.
  Incidence of Treatment Emergent Adverse Events (Study drugs: ciprofloxacin, 14C labelled ciprofloxacin and imipenem)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zeitlinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Oesterreicher Z, Eberl S, Wulkersdorfer B, Matzneller P, Eder C, van Duijn E, Vaes WHJ, Reiter B, Stimpfl T, Jager W, Nussbaumer-Proell A, Marhofer D, Marhofer P, Langer O, Zeitlinger M. Microdosing as a Potential Tool to Enhance Clinical Development of Novel Antibiotics: A Tissue and Plasma PK Feasibility Study with Ciprofloxacin. Clin Pharmacokinet. 2022 May;61(5):697-707. doi: 10.1007/s40262-021-01091-1. Epub 2022 Jan 7. PMID 34997559